CLINICAL TRIAL: NCT00447629
Title: A Randomized, Double-Blind, Placebo- and Moxifloxacin (Open-Label)- Controlled, 4-Period Crossover Study of the Effects of Single Oral Doses of PPM 204 on Cardiac Repolarization in Healthy Subjects
Brief Title: Study Evaluating Single Doses of PPM-204 on the Electrical Pathways of the Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3180A1-1109
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: PPM-204

SUMMARY:
A study evaluating the safety of a high and low dose of PPM-204 on the electrical pathways of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged 18 to 55 years
* Body mass index in the range of 18 to 30 kg/m2
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECG

Exclusion Criteria:

* History of cardiac, thyroid, muscle, or kidney abnormalities
* A family history of long QT syndrome and/or sudden cardiac death
* History of any clinically significant drug allergy, hypersensitivity to sulfonomides or the quinolone class of antibiotics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Phoenix, Arizona, United States